CLINICAL TRIAL: NCT06706297
Title: Effect of Breathıng Exercıse Applıed to Indıvıduals Wıth Copd on Respıratory Functıon, Dyspnea and Qualıty of Lıfe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Aybike Kose, Specialist Nurse,, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OMU-SBF-HEM-01
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life
Keywords: Dyspnea; COPD; Breathing Exercise; Pranayama; Respiratory Function; Quality of Life.
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This research was planned as a prospective, randomized controlled, experimental type study with pretest-posttest measurements to determine the effect of breathing exercise on dyspnea, respiratory function and quality of life in patients with COPD.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Control group patients will not undergo any exercise and the normal clinical protocol will not be interfered with.
- breathing exercise group (Experimental): The researcher will make the application group patients perform a 30-minute pranayama exercise twice a week for 6 weeks.
  Interventions: Other: pranayama breathing exercise

INTERVENTIONS:
Other: pranayama breathing exercise — Normal breathing, focusing on breathing, Alternative Nose Breathing, Cooling Breath, Bee Buzzing Sound, A breathing exercise of 20 minutes in total, consisting of 5 stages: normal breathing and focusing on breathing.
  Arms: breathing exercise group

SUMMARY:
Purpose of the research This research was designed to determine the effect of breathing exercise applied to individuals diagnosed with COPD on respiratory function, dyspnea and quality of life.

Hypotheses of the Research H0a: Breathing exercise applied to individuals diagnosed with COPD has no effect on the respiratory function test FEV1/FVC.

H1a: Breathing exercise applied to individuals diagnosed with COPD has an effect on the respiratory function test FEV1/FVC.

H0b: Breathing exercise applied to individuals diagnosed with COPD has no effect on dyspnea.

H1b: Breathing exercise applied to individuals diagnosed with COPD has an effect on dyspnea.

H0c: Breathing exercise applied to individuals diagnosed with COPD has no effect on quality of life.

H1c: Breathing exercise applied to individuals diagnosed with COPD has an effect on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD for at least 1 year, confirmed by pulmonary function test
* Those who voluntarily accepted to participate in the research
* Those aged 18 and over,
* Individuals who have access to the hospital

Exclusion Criteria:

* In COPD exacerbation period,
* Having a neurological or psychiatric diagnosis,
* Those with obesity,
* Those with physical disabilities (vision, hearing, walking, etc.),
* Those who are pregnant,
* Illiterate
* Diagnosed with another disease that significantly affects the respiratory system (scoliosis, lung cancer, abdominal tumor, etc.).
* Patients who have previously participated in an exercise program will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
pulmonary function test | 6 weeks
  The effect of breathing exercise applied to individuals with COPD on respiratory function test FEV1/FVC
Dyspnea severity | 6 weeks
  The effect of breathing exercise applied to individuals with COPD on dyspnea
Saint George's Solunum Anket | 6 weeks
  The effect of breathing exercise applied to individuals with COPD on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Aybike KÖSE, 1, Study Chair — Ondokuz Mayıs University; Afitap ÖZDELİKARA, 2, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No